CLINICAL TRIAL: NCT02241538
Title: Cost Effectiveness and Effectiveness of the Addition of Different Weekly Frequency of Modified Pilates Method Exercises to a Minimal Intervention in the Treatment of Chronic Nonspecific Low Back Pain: A Randomized Controlled Trial
Brief Title: Effectiveness of Different Weekly Frequency of Modified Pilates Method Exercises in the Treatment of Chronic Nonspecific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Cidade de Sao Paulo (Other)
Responsible Party: Principal Investigator, Cristina Maria Nunes Cabral, Associate Professor, Universidade Cidade de Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 29303014.7.0000.0064
Record Dates: First submitted 2014-09-12; First posted 2014-09-16 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Low Back Pain
Keywords: Pilates-based exercises
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Pilates 1 (Experimental): Combination of an educational booklet with exercises of the Pilates method. Patients will receive 6 sessions of treatment over a period of 6 weeks (1 session/week). The exercises of the Pilates method will be individualized to each patient´s needs (pragmatic treatment).
  Interventions: Device: Pilates 1
- Pilates 2 (Experimental): Combination of an educational booklet with exercises of the Pilates method. Patients will receive 12 sessions of treatment over a period of 6 weeks (2 sessions/week). The exercises of the Pilates method will be individualized to each patient´s needs (pragmatic treatment).
  Interventions: Device: Pilates 2
- Pilates 3 (Experimental): Combination of an educational booklet with exercises of the Pilates method. Patients will receive 18 sessions of treatment over a period of 6 weeks (3 sessions/week). The exercises of the Pilates method will be individualized to each patient´s needs (pragmatic treatment).
  Interventions: Device: Pilates 3
- Control (Active Comparator): Patients will receive an educational booklet containing information about the anatomy of the spine and pelvis and the low back pain and recommendations regarding posture and movements involved in activities of daily living. The participants in this group will not receive additional exercise.
  Interventions: Device: Control

INTERVENTIONS:
Device: Pilates 1 — Combination of an educational booklet with exercises of the Pilates method. Patients will receive 6 sessions of treatment over a period of 6 weeks (1 session/week). The exercises of the Pilates method will be individualized to each patient´s needs (pragmatic treatment).
  Arms: Pilates 1
Device: Pilates 2 — Combination of an educational booklet with exercises of the Pilates method. Patients will receive 12 sessions of treatment over a period of 6 weeks (2 sessions/week). The exercises of the Pilates method will be individualized to each patient´s needs (pragmatic treatment).
  Arms: Pilates 2
Device: Pilates 3 — Combination of an educational booklet with exercises of the Pilates method. Patients will receive 18 sessions of treatment over a period of 6 weeks (3 sessions/week). The exercises of the Pilates method will be individualized to each patient´s needs (pragmatic treatment).
  Arms: Pilates 3
Device: Control — Patients will receive an educational booklet containing information about the anatomy of the spine and pelvis and the low back pain and recommendations regarding posture and movements involved in activities of daily living. The participants in this group did not receive additional exercise.
  Arms: Control

SUMMARY:
Low back pain is a major cause of disability and absenteeism and the supervised exercise is a recommended treatment by the guidelines and has been cost-effective. Currently, the Pilates method has shown to be effective in improving pain and disability in patients with chronic low back pain (CLBP). However, there is still no evidence about the ideal number of sessions for the treatment and the interval between sessions to achieve better efficacy of this method for these patients. Thus, the aim of this study is to investigate the effectiveness of the Pilates method with different weekly frequency of sessions in the treatment of patients with nonspecific CLBP. Investigators will assess 296 patients of both genders, with nonspecific CLBP lasting more than three months and aged between 18 and 80 years. Participants will be randomly divided into four groups (n = 74 patients per group): Control Group will receive an educational booklet and no additional exercise, Pilates 1 Group will receive a program of exercises based on Pilates method once a week for six weeks, Pilates 2 Group will receive the same program of exercises twice a week for six weeks and Pilates 3 Group will receive the same program of exercises three times a week for six weeks. The outcomes overall disability (Roland Morris Disability questionnaire), specific disability (Patient-Specific Functional scale), kinesiophobia (Tampa scale for kinesiophobia), pain intensity (Pain Numerical Rating scale) and global perceived effect (Global Perceived Effect scale) will be assessed by a blinded assessor before, six weeks, six and 12 months after randomization. Investigators expect that the largest number of weekly sessions of Pilates method may influence the results in all analyzes (short, medium and long term), since there is a relationship between frequency of exercises and effect size of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic nonspecific low back pain longer 12 weeks

Exclusion Criteria:

* Contra indications to physical exercise
* Serious spinal pathologies (e. g. tumors, fractures and inflammatory diseases)
* Nerve root compromise
* Pregnancy
* Previous surgery on spine
* Pilates treatment for low back pain in the last three months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2014-09; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Six weeks after randomization
  Pain intensity will be measured by an 11-point Pain Numerical Rating Scale
Disability | Six weeks after randomization
  Disability associated with low back pain will be measured by the 24-item Roland Morris Disability Questionaire

SECONDARY OUTCOMES:
Pain intensity | Six and twelve months after randomization
  Pain intensity will be measured by an 11-point Pain Numerical Rating Scale
Disability | Six and twelve months after randomization
  Disability associated with low back pain will be measured by the 24-item Roland Morris Disability Questionaire
Global impression of recovery | Six weeks, six and twelve months after randomization
  Global impression of recovery will be measured by an 11-point Global Perceived Effect Scale
Specific disability | Six weeks, six and twelve months after randomizaion
  Specific disability will be evaluated by an 11-point Patient-specific Functional Scale
Kinesiophobia | Six weeks, six and twelve months after randomization
  Kinesiophobia will be evaluated by the Tampa Scale for Kinesiophobia
Pain-Related Catastrophizing | Six weeks, six and twelve months after randomization
  Pain-related catastrophizing will be evaluated by the Pain-Related Catastrophizing Thoughts Scale
Cost Effectiveness | Six weeks, six and twelve months after randomization
  Assessments of direct costs (patient out-of-pocket costs) by an specific questionnaire.
Quality Adjusted Life Years | Six weeks, six and twelve months after randomization
  Quality adjusted life years will be measured by the SF-6D questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Physical Therapy Outpatient Department, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Silva MLD, Miyamoto GC, Franco KFM, Franco YRDS, Cabral CMN. Different weekly frequencies of Pilates did not accelerate pain improvement in patients with chronic low back pain. Braz J Phys Ther. 2020 May-Jun;24(3):287-292. doi: 10.1016/j.bjpt.2019.05.001. Epub 2019 May 16. PMID 31153789
- [Derived] Miyamoto GC, Franco KFM, van Dongen JM, Franco YRDS, de Oliveira NTB, Amaral DDV, Branco ANC, da Silva ML, van Tulder MW, Cabral CMN. Different doses of Pilates-based exercise therapy for chronic low back pain: a randomised controlled trial with economic evaluation. Br J Sports Med. 2018 Jul;52(13):859-868. doi: 10.1136/bjsports-2017-098825. Epub 2018 Mar 10. PMID 29525763
- [Derived] Miyamoto GC, Moura KF, Franco YR, Oliveira NT, Amaral DD, Branco AN, Silva ML, Lin C, Cabral CM. Effectiveness and Cost-Effectiveness of Different Weekly Frequencies of Pilates for Chronic Low Back Pain: Randomized Controlled Trial. Phys Ther. 2016 Mar;96(3):382-9. doi: 10.2522/ptj.20150404. Epub 2015 Aug 20. PMID 26294680